CLINICAL TRIAL: NCT03545607
Title: MultiStem® Administration for Stroke Treatment and Enhanced Recovery Study (MASTERS-2)
Brief Title: MultiStem® Administration for Stroke Treatment and Enhanced Recovery Study
Acronym: MASTERS-2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Healios K.K. (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B01-04
Record Dates: First submitted 2018-05-23; First posted 2018-06-04 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; adult stem cells
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MultiStem (Experimental): 1.2 billion cells
  Interventions: Biological: MultiStem
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MultiStem — single intravenous infusion 18-36 hours after stroke
  Arms: MultiStem
Biological: Placebo — single intravenous infusion 18-36 hours after stroke
  Arms: Placebo

SUMMARY:
A Phase 3 study to examine the safety and effectiveness of the allogeneic, adult stem cell investigational product, MultiStem, in adults who have suffered an acute ischemic stroke in the previous 18-36 hours.

ELIGIBILITY:
Primary Inclusion Criteria:

* Male or female subjects ≥18 years of age
* Clinical diagnosis of ischemic stroke involving cerebral cortex
* Occurrence of a moderate to moderately severe stroke with a persistent neurologic deficit documented by a NIHSS score of 8 to 20 (inclusive) that does not change by ≥4 points during the initial screening period
* A mRS score of 0 or 1 prior to the onset of symptoms of the current stroke

Primary Exclusion Criteria:

* Presence of a lacunar or a brainstem infarct
* Comatose state
* Brain hemorrhage
* Major neurological event such as stroke or clinically significant head trauma within 6 months of enrollment into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-07-28 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
assessment of disability by examining the distribution of modified Rankin Scale (mRS) scores [scale range = 0 to 6] evaluated by shift analysis | 90 days

SECONDARY OUTCOMES:
proportion of subjects achieving an excellent functional outcome defined by all of the following criteria: | 365 days
  mRS score = 0 to 1 [scale range 0 to 6]; and NIHSS score = 0 to 1 [scale range 0 to 42]; and Barthel Index score = greater than or equal to 95 [scale range 0 to 100]
proportion of subjects achieving an excellent functional outcome defined by all of the following criteria: | 90 days
  mRS score = 0 to 1 [scale range 0 to 6]; and NIHSS score = 0 to 1 [scale range 0 to 42]; and Barthel Index score = greater than or equal to 95 [scale range 0 to 100]
proportion of subjects with a mRS score of less than or equal to 2 [scale range 0 to 6] demonstrating the ability to function independently | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Mays, PhD, Study Director — Healios K.K.
Locations (26):
- United States (23):
  - Athersys Investigational Site 128, Phoenix, Arizona
  - Athersys Investigational Site 122, Palo Alto, California
  - Athersys Investigational Site 127, Sacramento, California
  - Athersys Investigational Site 129, Clearwater, Florida
  - Athersys Investigational Site 108, Miami, Florida
  - Athersys Investigational Site 103, Augusta, Georgia
  - Athersys Investigational Site 121, Chicago, Illinois
  - Athersys Investigational Site 119, Kansas City, Kansas
  - Athersys Investigational Site 124, Wichita, Kansas
  - Athersys Investigational Site 113, Boston, Massachusetts
  - Athersys Investigational Site 125, Minneapolis, Minnesota
  - Athersys Investigational Site 111, Jackson, Mississippi
  - Athersys Investigational Site 109, Akron, Ohio
  - Athersys Investigational Site 104, Cleveland, Ohio
  - Athersys Investigational Site 130, Toledo, Ohio
  - Athersys Investigational Site 102, Portland, Oregon
  - Athersys Investigational Site 107, Hershey, Pennsylvania
  - Athersys Investigational Site 106, Pittsburgh, Pennsylvania
  - Athersys Investigational Site 118, Columbia, South Carolina
  - Athersys Investigational Site 115, Chattanooga, Tennessee
  - Athersys Investigational Site 101, Houston, Texas
  - Athersys Investigational Site 105, Houston, Texas
  - Athersys Investigational Site 110, Salt Lake City, Utah
- Taiwan (3):
  - Athersys Investigational Site 603, Taichung
  - Athersys Investigational Site 601, Taipei
  - Athersys Investigational Site 602, Taoyuan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hess DC, Wechsler LR, Clark WM, Savitz SI, Ford GA, Chiu D, Yavagal DR, Uchino K, Liebeskind DS, Auchus AP, Sen S, Sila CA, Vest JD, Mays RW. Safety and efficacy of multipotent adult progenitor cells in acute ischaemic stroke (MASTERS): a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Neurol. 2017 May;16(5):360-368. doi: 10.1016/S1474-4422(17)30046-7. Epub 2017 Mar 17. PMID 28320635